CLINICAL TRIAL: NCT00188344
Title: A Randomized Comparison of Laparoscopic Myotomy and Pneumatic Dilatation for Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT-76449; ISRCTN05714772
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Esophageal Achalasia
Keywords: laparoscopic myotomy; pneumatic dilatation; motility disorder; dysphasia; health-related quality of life
MeSH Terms: conditions — Esophageal Achalasia; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): pneumatic dilatation
  Interventions: Procedure: pneumatic dilatation
- 2 (Active Comparator): Laparoscopic myotomy
  Interventions: Procedure: laparoscopic myotomy with partial fundoplication

INTERVENTIONS:
Procedure: pneumatic dilatation — The patient is on a liquid diet for 2 days prior to procedure. A sedative and pain killer by IV are given and the throat will be sprayed with local anesthetic.
  The gastroenterologist may perform an endoscopy prior to the dilatation to safely guide the dilator into position. A special dilator with a small balloon will be passed down the esophagus until it meets the stomach then the balloon will be inflated with air until the narrow part of the esophagus is opened. The patient will then be assessed for any perforation of the esophagus and monitored in the post-procedure unit for a few hours.
  Arms: 1
Procedure: laparoscopic myotomy with partial fundoplication — The abdomen is inflated with gas and cameras and instruments are inserted. The junction between the esophagus and stomach is identified. The muscle of the lower esophageal sphincter is divided. A portion of the stomach wall is secured to the lower esophagus. After surgery the patient is taken to the recovery room and when well enough moved to a ward. The patient may be discharged the following day.
  Arms: 2

SUMMARY:
The purpose of this study is to compare pneumatic dilatation and laparoscopic Heller myotomy in patients with achalasia in order to learn which of these two treatments should be recommended to patients in the future.

DETAILED DESCRIPTION:
Achalasia is a rare disease of the esophagus. It can cause difficulty swallowing, regurgitation of swallowed food, and chest pain. In achalasia, there are two problems in the esophagus. First, the esophagus does not properly push swallowed food down towards the stomach. Second, the valve at the lower end of the esophagus, called the lower esophageal sphincter, does not relax to allow food to pass from the esophagus into the stomach.

Achalasia cannot be "cured". However, the symptoms of achalasia can be improved by treatment. Treatment is usually directed towards reducing the degree of blockage caused by the lower esophageal sphincter. the muscle of the lower esophageal sphincter can be stretched using a technique called pneumatic dilatation, or it can be divided (cut in half) during a surgical operation. The operation is called laparoscopic Heller myotomy, and is done by laparoscopic ("keyhole") surgery, where small incisions are used and patients usually stay in hospital 1-2 nights. Other treatments for achalasia, such as medications or injection of Botulinum Toxin Type A are not often used because they do not provide effective long-term improvement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of achalasia by a physician
* manometric diagnosis of achalasia including both: Incomplete relaxation of the lower esophageal sphincter during swallowing (<80% of elevation over intragastric pressure and absence of esophageal peristalsis (peristalsis in <20% of initiated contractions)
* Facility with English, ability to complete English language questionnaires

Exclusion Criteria:

* Pseudoachalasia: esophageal carcinoma; esophageal stricture; previous esophageal or gastric surgery; previous instrumentation of the lower esophageal sphincter i.e. suture, polymer injection, silicone band
* Previous gastric or esophageal surgery: fundoplication; Heller myotomy; gastric resection; vagotomy with or without gastric drainage
* Age 17 year or less
* Pregnancy
* Presence of severe comorbid illness: unstable angina; recent myocardial infarction (<6 months), cancer (except integumentary), unless free of disease for more than 5 years; end stage renal disease; previous stroke with cognitive, motor speech, or swallowing deficit persisting longer than one month; severe respiratory disease; cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The achalasia severity questionnaire score at 1 year. | Baseline, M2, M6, Yrs 1 to 5

SECONDARY OUTCOMES:
Generic health related quality of life (SF-36) | baseline, M2, M6, Yrs 1 to 5
Gastrointestinal disease-specific quality of life (GIQLI) | baseline, M2, M6, Yrs 1 to 5
Measures of esophageal physiology | baseline, M6
Gastroesophageal reflux as measured by ambulatory 24-hr esophageal pH measurement | M6
Clinical outcomes of care including short term outcomes, major complications, and long-term clinical outcomes. | Yrs 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: David R Urbach, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, 30 Bond Street, Suite 16 048 Cardinal Carter Wing, Toronto, Ontario
  - University Health Network, Toronto, Ontario